CLINICAL TRIAL: NCT02106754
Title: Alcohol Screening & Brief Lntervention in Juvenile Justice: Filling the Gap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Lynda Stein, Ph.D., Professor, University of Rhode Island, University of Rhode Island
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R01AA021855 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-08 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Evaluating NIAAA's Alcohol Screener; Evaluating a Brief Intervention
MeSH Terms: interventions — Crisis Intervention; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Intervention (Experimental): Youth may receive brief intervention from their provider based on randomization.
  Interventions: Behavioral: Brief Intervention
- Treatment As Usual (Active Comparator): Youth may receive treatment as usual from their provider based on randomization.
  Interventions: Behavioral: Treatment as Usual
- Brief Intervention with Coaching (Experimental): Youth may receive brief intervention with coaching from their provider based on randomization.
  Interventions: Behavioral: Brief Intervention with Coaching

INTERVENTIONS:
Behavioral: Brief Intervention
  Arms: Brief Intervention
Behavioral: Brief Intervention with Coaching
  Arms: Brief Intervention with Coaching
Behavioral: Treatment as Usual
  Arms: Treatment As Usual

SUMMARY:
This proposal is in response to RFA-AA-12-008, Evaluation of NIAAA's Alcohol Screening Guide for Children and Adolescents. Of particular interest to the agency are evaluation of the Screener in clinical and/or other settings to predict alcohol-related consequences including use disorder; its use as an initial screen for drug use, cigarette smoking, conduct disorder, and unprotected sex; and its performance in making predictions concurrently and prospectively. This proposal targets these areas of interest. In addition, the investigators will study implementation of the Brief Intervention (BI) associated with the Screener. There is a great need for both screening and BI in juvenile probation settings as many of these youths have great need but are underserved.Many probation departments are turning to BI to work with probationers and parolees. Screening and BI has demonstrated efficacy in these settings, and yet no randomized control trials have been conducted to evaluate effectiveness in juvenile probation settings. Probation Officers (POs; n=40) are randomized to Screener (S), Screener+BI (SBI), or coaching (CSBI). Youths (N=1000) are randomized to 1 of these 3 conditions, and all receive usual services (US). US consist of regular check-in with PO and access to referral services as needed (counseling, academic tutoring, etc.). Research staffers conduct in-depth assessment at baseline, 6- and 12- months. Sensitivity, specificity, and positive and negative predictive powers (SN, SP, PP, NP) are calculated to predict alcohol risk and consequences, as well as other risky behaviors concurrently and prospectively across age-groups. A 1-way design (S vs SBI vs CSBI) will be used to determine whether SBI and CSBI enhance youth services-use and reduce risks (e.g., alcohol use, risky sex). We examine moderators of outcomes (youth age, PO characteristics) and whether coaching (an important consideration in implementation science) in use of BI improves outcomes. This study will be the first randomized controlled trial evaluating the effectiveness of SBI in a juvenile probation setting.

DETAILED DESCRIPTION:
1. A) To evaluate SN, SP, PP and NP of the 2-question Alcohol Screener to detect: a) alcohol problems (academic, social, injuries, intoxicated driving, unprotected sex), b) abuse/dependence, c) past 4 week binge drinking. 1B) This will be repeated to predict risk prospectively over 12 months. Classification rates will be compared for race, ethnicity, gender, and age groups.
2. A) To evaluate SN, SP, PP and NP of the 2-question Screener to detect a) 30-day drug use, b) 30-day cigarette use, c) conduct disorder, d) unprotected sex. 2B) This will be repeated to predict risk prospectively over 12 months. Classification rates will be compared for race, ethnicity, gender, and age groups. 3) To evaluate BI as compared to usual procedures. The investigators hypothesize those youths in BI will a) receive more services, b) be more satisfied with services, c) rate the relationship with the PO more highly, and d) have improved outcomes (alcohol, alcohol-related problems, problem recognition).

ELIGIBILITY:
Inclusion Criteria:

* Youths 9-18 years old

Exclusion Criteria:

* Age (< 9, >18 years)
* Prior enrollment in a behavioral intervention study
* PO previously engaging them with Screener

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 576 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Measure of change across three points in time for alcohol, cigarette and other drug use | baseline, 6 month follow-up, 12 month follow-up
  Time-Line Follow-Back (TLFB) measures past 30-day use of alcohol, cigarettes, and other drugs at each assessment (BL, 6- & 12-month). It is well known, reliable and valid (Harrison & McKee, 2008; Carey et al, 2004). Days/month used, and binge-drinking are obtained. For analyses involving classification rates, binge >
  1 is considered problematic, and definitions of binge will follow Donovan (2009).
  RCQ (Risks/Consequences Questionnaire; Stein et al, 2010) provides an overall

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Stein, Principal Investigator — URI
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No